CLINICAL TRIAL: NCT01954069
Title: Simplifying Menstrual Regulation (MR): Exploring the Role of At-home Semi-quantitative Pregnancy Tests for Follow-up to Menstrual Regulation Service Provision in Pakistan
Brief Title: Exploring the Role of At-home Semi-quantitative Pregnancy Tests for Follow-up to Menstrual Regulation Service
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 6005
Record Dates: First submitted 2013-09-26; First posted 2013-10-01 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: Menstrual Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Semi-quantitative pregnancy test (Other): Semi-quantitative urine pregnancy test (SQPT) (dBest One Step hCG Panel Test Kit)
  Interventions: Device: Semi-quantitative pregnancy test

INTERVENTIONS:
Device: Semi-quantitative pregnancy test
  Other Names: semi-quantitative urine pregnancy test (SQPT) (dBest One Step hCG Panel Test Kit)

SUMMARY:
The study seeks to test whether it is feasible and acceptable for both women and providers (in this context the Lady Health Visitor) to use the semi-quantitative pregnancy test (SQPT) as a tool for follow up after MR services. The study is planned at 11service delivery points (primary health clinics) in Punjab province where consenting women will be asked to take a baseline test at the clinic the morning they present for the MR procedure. Women will be asked to complete a second test at home the morning of their scheduled follow up visit and return to the clinic for follow-up care later that day. The results of the at home test will be compared to the baseline to determine the outcome of the MR. This is of particular importance because to-date no research has documented the accuracy of the test in detecting MR outcomes with misoprostol only regimens.

We hypothesize that women and providers will find the test easy and acceptable to use thereby improving follow up and simplifying MR service provision. In addition, the simple pictorial instructions will enable most women to use the test and interpret the results correctly on their own.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for medical menstrual regulation services according to clinic guidelines
* Willing to follow instructions and use the SQPT at home
* Agrees to return for a follow-up visit 7 days after receipt of misoprostol for the MR procedure

Exclusion Criteria:

* Not eligible for medical menstrual regulation services according to clinic guidelines
* Not willing to follow instructions and use the SQPT at home
* Does not agree to return for a follow-up visit 7 days after receipt of misoprostol for the MR procedure

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2013-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Feasibility to determine successful completion of MR | 2 weeks
  1. The proportion of woman for whom Human Chorionic Gonadotropin (hCG) remains the same after MR
  2. The proportion of woman for whom hCG remains increases after MR
  3. The proportion of woman for whom hCG declines after MR
  4. Any additional care received by women in each of the above groups (1-3) will also be described

SECONDARY OUTCOMES:
Comprehension of pregnancy test | 2 weeks
  Proportion of women who correctly read and interpreted their results
Confidence in test | 2 weeks
  Proportion of women who were confident in using the test and would be willing to use it for follow up in the future
Selecting and receiving family planning method | 2 weeks
  Proportion of women selecting a method of family planning and receiving that method at their initial clinic visit.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Blum, MPH, Principal Investigator — Gynuity Health Projects; Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects; Asifa Khanum, MPhil, MSc, Principal Investigator — Rahnuma FPAP; Anjum Rizvi, MBBS, MHA, Principal Investigator — Rahnuma FPAP; Dina Abbas, MPH, Principal Investigator — Gynuity Health Projects
Locations (11):
- Pakistan (11):
  - Bhagwal Service Delivery Clinic, Bhagwal, Chakwal
  - Chakumra Service Delivery Clinic, Chakumra, Chakwal
  - Karrila Service Delivery Clinic, Karrila, Chakwal
  - Khanpur Service Delivery Clinic, Khanpur, Chakwal
  - Chak 128 GB Service Delivery Clinic, Faisalabad, Faisalabad
  - BagaSher Service Delivery Clinic, BagaSher, Muzaffargarh
  - Dasrat Colony Service Delivery Clinic, Dasrat Colony, Muzaffargarh
  - Fazal Nagal Service Delivery Clinic, Fazal Nagal, Muzaffargarh
  - TibbiAryain Service Delivery Clinic, TibbiAryain, Muzaffargarh
  - Bahari Colony Service Delivery Clinic, Bahari Colony, Rawalpindi
  - DhokeHasso Service Delivery Clinic, DhokeHasso, Rawalpindi